CLINICAL TRIAL: NCT05073887
Title: A Comparison of Ultrasound Guided Genicular Nerve Blockade Using Current Versus Revised Anatomical Targets in Chronic Knee Osteoarthritis: A Double-Blind, Randomized Controlled Trial
Brief Title: A Comparison of Ultrasound Guided Genicular Nerve Blockade Using Current Versus Revised Anatomical Targets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Selin Guven Kose, principal investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 106/01
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Knee Pain Chronic
Keywords: Osteoarthritis; Radiofrequency; Ultrasound; Anatomical landmarks
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 nerve (Experimental): 3 genicular nerve blockade and radio frequency ablation
  Interventions: Procedure: Current Targets
- 5 nerve (Active Comparator): 3 genicular nerve blockade and radio frequency ablation 2 genicular nerve blockade and pulse radio frequency
  Interventions: Procedure: Current Targets

INTERVENTIONS:
Procedure: Current Targets — blockade and radio frequency stimulation of genicular nerves
  Other Names: Revised Targets

SUMMARY:
comparison of effectiveness of ultrasound guided genicular nerve blockades and radio frequency stimulation

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Coagulation disorders
* Rheumatoid disorders
* Infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale | Post injection sixth month
  Pain will be evaluated with a Numerical Rating Scale (NRS) score of 0-10 (0= no pain and 10= worst imaginable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Selin Guven Kose, Principal Investigator — Diskapi Yildirim Beyazit Education and Research Hospital
Locations (1):
- Diskapi Yildirim Beyazit Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guven Kose S, Kirac Unal Z, Kose HC, Celikel F, Akkaya OT. Ultrasound-guided genicular nerve radiofrequency treatment: prospective randomized comparative trial of a 3-nerve protocol versus a 5-nerve protocol. Pain Med. 2023 Jul 5;24(7):758-767. doi: 10.1093/pm/pnad025. PMID 36869680